CLINICAL TRIAL: NCT02242565
Title: Safety and Effectiveness of Different ShangRing Device Sizes for Adult Male Circumcision in Lusaka, Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Ministry of Health, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 576424; 010-04-14 (Other: UNZABREC (local IRB))
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Male Circumcision
Keywords: HIV prevention; ShangRing; adverse events; wound healing; voluntary medical male circumcision (VMMC); medical device; Zambia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: all-sizes of ShangRing (Other): All-sizes of ShangRings will be available.
  Interventions: Device: ShangRing
- Reduced-sizes (Active Comparator): 7 adult sizes of ShangRings will be available
  Interventions: Device: ShangRing

INTERVENTIONS:
Device: ShangRing — ShangRing device for male circumcision

SUMMARY:
The purpose of this study was to assess the safety, effectiveness and acceptability of providing a reduced number of ShangRing sizes for adult voluntary medical male circumcision (VMMC) within routine service delivery in Lusaka, Zambia.

DETAILED DESCRIPTION:
We conducted a randomized controlled trial and enrolled 500 HIV-negative men aged 18-49 years at 3 clinics. Participants were randomized to 1 of 2 study arms (Standard Sizing arm vs Modified Sizing arm) in a 1:1 ratio. All 14 adult ShangRing sizes (40-26 mm inner diameter, each varying by 1 mm) were available in the Standard Sizing arm; the Modified Sizing arm used every other size (40, 38, 36, 34, 32, 30, 28 mm inner diameter). Each participant was scheduled for 2 follow-up visits: the removal visit (day 7 after placement) and the healing check visit (day 42 after placement), when they were evaluated for adverse events (AEs), pain, and healing.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 to 49 years;
* Must be HIV-uninfected per same-day routine voluntary testing at the clinic;
* Must be uncircumcised (on examination);
* Must be in good general health, at the discretion of the clinician;
* Must be free of genital ulcerations or other visible signs of STI (on examination);
* Must be able to understand study procedures, and agree to abide by them including the follow-up visit schedule;
* Must freely consent to participate in the study and sign a written informed consent form;
* Must provide full contact information including cell phone number, address, and other locator information.

Exclusion Criteria:

* Has an active genital infection upon visual inspection;
* Has an anatomic abnormality (e.g. phimosis or hypospadias) that contraindicates ShangRing MMC;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid; or
* Has a self-reported medical condition that would be a contraindication for elective surgery, e.g. hemophilia, extreme obesity, poorly controlled diabetes, sickle cell anemia
* Has a self-reported allergy or sensitivity to lidocaine or other local
* Is not available to be circumcised on the same day as screening.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage and 95% confidence interval of men with at least one moderate or severe adverse event. | 42 days
  To assess the safety of ShangRing procedures when providers choose among 7 adult sizes (reduced-sizes or treatment arm) versus the full range of 14 adult sizes (all-sizes or control arm) during routine service delivery in Lusaka, Zambia.

SECONDARY OUTCOMES:
Percentage of men who cannot be properly fitted with a ShangRing device | 42 days
  Assess the effectiveness of ShangRing procedures in the reduced-sizes arm.
Evaluate the acceptability of ShangRing procedures among participants and providers | 42 days
  Participant acceptability (with procedure and cosmetic appearance), pain, and time to return to normal activity after ShangRing circumcision, overall and in each arm.
  Provider acceptability assessing ease, duration, and complications, and preferences comparing ShangRing with other methods of circumcision, and comparing reduced-sizes with all-sizes provision.
Percentage of men with complete healing at 42 days | Day 42
  Percentage of men with complete healing at 42 days for all study participants, and within each arm of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zulu, MD, Principal Investigator — University Teaching Hospital; Paul Feldblum, PhD, Principal Investigator — FHI 360
Locations (2):
- Zambia (2):
  - Chilenje Urban Health Centre, Lusaka
  - The University Teaching Hospital (UTH), Lusaka

REFERENCES:
- [Result] Feldblum PJ, Zulu R, Linyama D, Long S, Nonde TJ, Lai JJ, Kashitala J, Veena V, Kasonde P. Randomized Controlled Trial of the ShangRing for Adult Medical Male Circumcision: Safety, Effectiveness, and Acceptability of Using 7 Versus 14 Device Sizes. J Acquir Immune Defic Syndr. 2016 Jun 1;72 Suppl 1(Suppl 1):S30-5. doi: 10.1097/QAI.0000000000001015. PMID 27331587